CLINICAL TRIAL: NCT04191655
Title: High Definition Colonoscopy (HDC) vs. Dye Spraying Chromo-colonoscopy (DSC) in Screening Patients With Long-standing Inflammatory Bowel Disease (IBD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Feuerstein, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2018P000795
Record Dates: First submitted 2019-12-02; First posted 2019-12-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases; Colon Dysplasia; Ulcerative Colitis; Crohn Colitis; Indeterminate Colitis
Keywords: Colorectal cancer screening; Inflammatory bowel disease; Chromocolonoscopy; High definition white light colonoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Intervention Model Description: After patients consent to participate to the study, they will be randomized 1:1 by one of the study members who is blinded to the patient's history to either High Definition White Light Colonoscopy with biopsies every 10 cm or Dye Spraying Chromocolonoscopy. The gastroenterologist will be informed about the randomization result and s/he will conduct the procedure.
Who Masked: Participant, Care Provider, Investigator
Masking Description: In this study, we will randomize a total of 500 participants into two arms: A. high definition white light colonoscopy with biopsy (n=250) or B. chromocolonoscopy (n=250).
  The randomization schedule was created by using GraphPad website. Then sealed opaque envelopes which numbered from 1 to 500 for all subjects were created based on the randomization schedules by one of the study co-investigators (Mohammed El-Dallal MD). These envelopes will be opened only by the endoscopy provider once the subject agrees and sings the informed consent. Of note, the randomization schedules will be saved in a separate document that only Mohammed El-Dallal MD has access to it. Neither the participants nor the study members (other than Mohammed El-Dallal MD) know about the assignment before opening the envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Definition White Light Colonoscopy (Experimental)
  Interventions: Device: High Definition Colonoscopy
- Dye Spraying Chromo-colonoscopy (Active Comparator)
  Interventions: Device: Dye Spraying Chromocolonoscopy

INTERVENTIONS:
Device: High Definition Colonoscopy — A colonoscopy that used high definition (HD) camera
  Arms: High Definition White Light Colonoscopy
Device: Dye Spraying Chromocolonoscopy — A colonoscopy that used high definition camera in addition to dye spraying on the interior colon surface.
  Arms: Dye Spraying Chromo-colonoscopy

SUMMARY:
Inflammatory Bowel Disease (IBD) involving the colon is a known risk for colon cancer. There are two standards-of-care colonoscopy techniques used for screening all patients who suffer from IBD for more than eight years. One method is to obtain random biopsies throughout the colon and the other is by using dye spraying chromo-colonoscopy.

This trial aims to study the difference between the two colonoscopy techniques during the era of high definition camera in detecting neoplastic lesions during screening patients with long-standing IBD.

DETAILED DESCRIPTION:
Research Question:

Is High Definition White Light Colonoscopy (HDWLC) not inferior to Dye Spraying Chromo-colonoscopy (DSC) in detecting all neoplastic lesions during screening patients with colonic IBD for more than eight years?

Study setting: The study will be conducted at Beth Israel Deaconess Medical Center. Patients will be randomized to HDWLC with biopsies every 10 cm versus DSC.

Study population: Adult patients colonic IBD for more than eight years.

Recruitment The study team will conduct a day by day chart review for all patients with a history of inflammatory bowel disease who were scheduled for screening colonoscopy and find candidates who meet the eligibility criteria. A study team member will meet with the potential candidates during their visit to the gastroenterology procedure room before having their colonoscopy and offer them to participate in the study.

Procedures: Participants will undergo either HDWLC with biopsies every 10 cm or DSC based on the randomization. Both procedures are standard of care and are being done at BIDMC before starting this study. All the endoscopists are IBD specialists with expertise in both procedures. All physicians were given a review article and video of chromoendoscopy to further standardize practice. The clinicians who are conducting the HDWLC are allowed to do a targeted DSC if required as per hospital protocol. Both arms of the study are using high definition Olympus colonoscopes

Study design: A randomized controlled, noninferiority trial.

Sample size:

Existing literatures suggest that the detection rate of the DSC arm is 20%. The investigators set 10% as the non-inferiority margin. With a total of 400 subjects (200 in each arm), the study will have 80% power to detect non-inferiority with the type I error rate controlled at 0.05. To account for a potential 25% data attribution, the study team will enroll 500 subjects.

Statistical Analysis:

The baseline characteristics of the two trial arms will first be tabulated for potential imbalance in variables. Continuous variables will be summarized by typical parameters such as mean, standard deviation and range and compared using two-sample T-test (if the normality assumption holds) or Wilcoxon rank-sum test (if the normality assumption does not hold). Normality of distribution will be determined using the Kolmogorov-Smirnov goodness-of-fit test. Categorical data will be summarized by frequency and percentage and analyzed using the Chi-square or Fishers exact test, as appropriate.

The primary outcome will be compared using Z-test based on normal approximation of the sample proportions.

Outcome analysis:

Primary outcome analysis: Intention to treat Secondary outcome analysis: Per protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥18yr old
2. History of UC or colonic Crohn's disease or unclassified colitis patients with or without colonic adenoma history
3. Duration of ≥ eight years since diagnosis, or any duration with a diagnosis of primary sclerosing cholangitis
4. Mucosal lesion involves ≥ 1/3 of the colon

Exclusion Criteria:

1. History of colorectal cancer
2. History of total colectomy
3. Prior colonoscopy within the last 6 months
4. Allergy to dye spray
5. Poor bowel preparation
6. Unable to provide informed consent
7. Severe inflammation preventing visualization of the mucosa during the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of dysplastic lesions in High Definition White Light Colonoscopy versus Dye Spraying Chromo-colonoscopy | Immediately after the procedure

SECONDARY OUTCOMES:
Detection rate of Adenoma in both groups. | Immediately after the procedure
Detection rate of high-grade dysplasia in both groups. | Immediately after the procedure
Numbers of detected adenomas per patient. | Immediately after the procedure
Difference in withdrawal time to perform the procedure in both groups. | Immediately after the procedure
Difference in adverse event, mild (e.g.; nausea, vomiting, or abdominal pain that necessitate phone call from the patient to the provider, or sever (e.g.; GI bleeding, perforation, hospitalization after the procedure) for each arm. | Within one week from the procedure date
Number of targeted chromoendoscopies | Immediately after the procedure
Appropriateness of reported follow up recommendations per standard guideline recommendations | Immediately after the procedure

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts